CLINICAL TRIAL: NCT03320577
Title: Take a Deep Breath: Randomized Controlled Trial of the Effects of Breathing Exercises on Blood Pressure
Brief Title: Pranayama Breathing and Uncontrolled Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jane McElroy, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005875
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Class instruction of breathing exercises (Active Comparator): Class participation/instruction weekly for 6 weeks and requested to practice Pranayama breathing exercises of 15 minute duration for an additional 4x during the week; completed log that indicated time/date/duration of practice; weekly blood pressure measurements and turn in logs; week 10 and week 18 blood pressure measurements also obtained. Survey instruments completed at baseline, week 6, 10, 18.
  Interventions: Behavioral: Class instruction of breathing exercises
- DVD instruction of breathing exercises (Active Comparator): Received DVD with instructions and 15 minute Pranayama breathing exercises of 15 minute duration. Participants requested to practice breathing exercises 5x during the week for 6 week intervention; completed log that indicated time/date/duration of practice; weekly blood pressure measurements and turn in logs; week 10 and week 18 blood pressure measurements also obtained. Survey instruments completed at baseline, week 6, 10, 18.
  Interventions: Behavioral: DVD instruction of breathing exercises
- Control (Placebo Comparator): Completed log that indicated time of eating dinner; weekly blood pressure measurements for the 6 week intervention; control participants also turned in dinner time logs; week 10 and week 18 blood pressure measurements also obtained. Survey instruments completed at baseline, week 6, 10, 18.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Class instruction of breathing exercises — Pranayama Breathing exercises practiced at least 5 times a week and log practice times
  Arms: Class instruction of breathing exercises
Behavioral: DVD instruction of breathing exercises — Pranayama Breathing exercises practiced at least 5 times a week and log practice times
  Arms: DVD instruction of breathing exercises
Behavioral: Control — Log dinner times
  Arms: Control

SUMMARY:
This study will compare participants who have uncontrolled hypertension and perform a set of five breathing exercises (Pranayama breathing) to a control group. The purpose of the study is to determine the effect of the breathing exercises on reduction of blood pressure.

DETAILED DESCRIPTION:
Untreated or uncontrolled hypertension is a leading cause of heart disease, stroke, and kidney failure. Hypertension, is a modifiable risk factor that may be successfully treated using one or a combination of treatment options, including medication, diet, exercise, tobacco cessation, or complementary and alternative medicine such as breathing exercises. A well-established cascade of adverse health outcomes are associated with hypertension as well as increased mortality rates. For patient-centered care, providing patients with additional strategies for their health care also has the potential to empower the patient, augment patient-physician team approach to the patient's health care, and support the standards of care for treating hypertension. As explained by McCaffrey et al from their focus group work with patients, "Participants do not want prescription medications except as a last resort and feel that conventional medicine overemphasizes prescription medicines. This may be because of a combination of factors including distrust in conventional medicine, fear of side effects from medicines, and an underlying belief that the body can heal itself given the right nutrition, rest, and time"

Using a randomized controlled trial study design with a 1-month and 3-month follow-up, the investigators hypothesize that practicing breathing at least 5 times per week will show a mean reduction in systolic (SBP) and diastolic (DBP) blood pressures in uncontrolled hypertensive patients compared to control patients. Participants will be randomized into one of three arms of the study. For the intervention arm, participants will be either assigned to a weekly class for the pranayama breathing instruction and practice or given a DVD that contains instructions on the breathing exercises and the 15-minute practice session.

ELIGIBILITY:
Inclusion Criteria

* English-speaking adults
* less than 60 years of age with BP measurements of ≥140/ ≥90 mm Hg
* 60 years of age or older with BP measurements of ≥150/ ≥90 mm Hg
* diagnosed with diabetes with BP measurements of ≥140/ ≥90 mm Hg
* Patients with BP measurements of <180/ <110 mm Hg without hypertensive urgency symptoms

Exclusion Criteria:

comorbidities of COPD, renal disease or chronic alcoholism

-

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Reduced blood pressure from breathing exercises | Baseline to week 10
  5 mmHg point reduction in blood pressure (dichotomous variable) associated with breathing exercises

SECONDARY OUTCOMES:
Beta blocker medication affect on blood pressure reduction | Baseline to week 6
  Differences on blood pressure (mean mmHg) reduction stratified by use of beta blockers (dichotomous)
Perceived political stress level of participant affect on blood pressure reduction | Baseline to week 10
  Differences on blood pressure (mean mmHg / dichotomous 5 mmHg reduction) reduction stratified by participants reported stress using one question about stress related to the 2016 elelction rated on a 5-point Likert scale from high stress (extremely-somewhat) to low stress (slightly-not at all); range 5-1;
Self Efficacy response to breathing exercises | Baseline to week 18
  General self efficacy scale ( point change; range: 10-40) increase in response to breathing exercises
Depressive severity response to breathing exercises | Baseline to week 18
  % participants who had PHQ-9 Patient Health Questionnaire which screens for depression (score <5 or >9; range 0-27) in response to breathing exercises

CONTACTS AND LOCATIONS:
Overall Officials: Jane A McElroy, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No